CLINICAL TRIAL: NCT05523869
Title: A Prospective Matched Cohort Study of Intravitreal Topotecan in the Repair of Rhegmatogenous Retinal Detachment with Proliferative Vitreoretinopathy
Brief Title: Intravitreal Topotecan in the Repair of Rhegmatogenous Retinal Detachment with Proliferative Vitreoretinopathy
Acronym: TOPO-RD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOPO-RD
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Proliferative Vitreoretinopathy in Rhegmatogenous Retinal Detachment
MeSH Terms: interventions — Scleral Buckling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravitreal topotecan with pars plana vitrectomy with or without scleral buckle (Experimental)
  Interventions: Drug: Intravitreal topotecan; Procedure: Pars plana vitrectomy with or without scleral buckle
- Pars plana vitrectomy with or without scleral buckle (Active Comparator)
  Interventions: Procedure: Pars plana vitrectomy with or without scleral buckle

INTERVENTIONS:
Drug: Intravitreal topotecan — Patients meeting all inclusion criteria and not meeting exclusion criteria will be assigned to receive pars plana vitrectomy with or without scleral buckle with intravitreal topotecan 8 µg/0.1mL, administered preoperatively within one week from surgery, intraoperatively during surgery, as well as postoperatively at 2 weeks, 4 weeks, 8 weeks, 12 weeks and 16 weeks, for a total of 7 injections.
  Arms: Intravitreal topotecan with pars plana vitrectomy with or without scleral buckle
Procedure: Pars plana vitrectomy with or without scleral buckle — Standard three-port pars plana vitrectomy with or without scleral buckle.

SUMMARY:
Intravitreal topotecan has anti-inflammatory, anti-proliferative and anti-fibrotic activity that we hypothesize may exhibit high efficacy for the treatment of proliferative vitreoretinopathy (PVR) in patients with rhegmatogenous retinal detachment (RRD). A high efficacy for intravitreal topotecan has been exhibited in cell cultures of PVR. At the same time, intravitreal topotecan has been routinely used in the treatment of vitreous seeds from retinoblastoma. At doses of 5-30 micrograms per injection, no adverse events have been reported with the use of intravitreal topotecan. Therefore, the current prospective matched phase II trial aims to investigate the efficacy and safety of intravitreal topotecan for severe PVR in patients with RRD.

ELIGIBILITY:
To be enrolled, patients need to meet the following inclusion criteria:

1. patients aged 18 years and older
2. patients who undergo PPV and/or SB for recurrent RRD due to PVR
3. patients with RRD and PVR grade C or D
4. patients who have failed standard of care surgery for RRD in the same eye previously. In order to satisfy this inclusion criterion, patients need to have previously received at least one vitreoretinal surgery for RRD, including pneumatic retinopexy, pars plana vitrectomy and/or scleral buckle, and to have clinical documentation supporting re-detachment of the retina after one or more vitreoretinal surgeries for RRD in the same eye. This cohort of patients is expected to have an extremely guarded visual prognosis and visual potential.
5. patients who are voluntarily able and willing to participate Patients undergoing combined phacoemulsification and PPV and/or SB will also be included. Any surgical technique will be considered, including relaxing retinotomy or retinectomy during PPV.

The following subject exclusion criteria will be considered:

1. patients with a history of tractional or exudative retinal detachment
2. patients with severe non-proliferative or proliferative diabetic retinopathy
3. patients with other planned ocular surgery following PPV
4. patients with primary RRD
5. female patients of childbearing age (i.e. less than 50 years old).
6. patients with pre-existing bone marrow suppression or cytopenias
7. patients with pre-existing interstitial lung disease (ILD) Any other medications or treatments, including rescue therapy, will be permitted before and/or during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Recurrent RRD secondary to PVR | 6 months or last follow-up

SECONDARY OUTCOMES:
Best corrected visual acuity | 6 months or last follow-up
Proliferative vitreoretinopathy grade | 6 months or last follow-up
Retinal reattachment rate | 6 months or last follow-up
Complications | 6 months or last follow-up
Best corrected visual acuity change from baseline | 6 months or last follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No